CLINICAL TRIAL: NCT01273389
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Proof-of-Concept Study to Evaluate Efficacy and Safety of Treatment With CNTO 136 Administered Intravenously in Subjects With Active Lupus Nephritis
Brief Title: An Efficacy and Safety Study of CNTO 136 in Patients With Active Lupus Nephritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR017551; CNTO136LUN2001 (Other: Janssen Research & Development, LLC); 2010-020968-38 (EudraCT Number); NCT01634581 (obsolete NCT alias)
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-02

CONDITIONS: Lupus Nephritis
Keywords: Lupus nephritis; CNTO 136; Sirukumab; Kidney diseases; Proteinuria; Glomerulonephritis
MeSH Terms: conditions — Lupus Nephritis; Kidney Diseases; Proteinuria; Glomerulonephritis | interventions — sirukumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CNTO 136 (Experimental): CNTO 136 is used in the form of final vialed product, as a single-use, sterile solution in a 2 ml glass vial. Each 1 mL of the solution contains sirukumab 100mg active drug substance, sorbitol, acetate buffer, and polysorbate 20, at a pH of 5.0, without any preservatives.
  Interventions: Drug: CNTO 136
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CNTO 136 — Type=exact number, unit=mg/kg, number=10, form=solution for injection, route=intravenous. CNTO 136 is administered once every 4 weeks from Week 0 to Week 24.
  Arms: CNTO 136
Drug: Placebo — Form=solution for injection, route=intravenous. Placebo is administered once every 4 weeks from Week 0 to Week 24.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of CNTO 136 administered intravenously in patients with active, International Society of Nephrology/Renal Pathology Society Class III and IV Lupus Nephritis (LN).

DETAILED DESCRIPTION:
This is a multicenter (study conducted at multiple sites), randomized (the study medication is assigned by chance), double-blind (neither investigator nor the patient knows the treatment that the patient receives), placebo-controlled (an inactive substance that is compared with the study medication to test whether the study medication has a real effect in clinical study), parallel group (each group of patients will be treated at the same time) study of CNTO 136 in patients with active LN. The study consists of 3 phases, ie, the screening phase (approximately 8 weeks prior randomization), treatment phase (24 weeks), and the follow up phase (through week 40). An 8 week run-in period will be used to establish the stability of baseline renal parameters prior to randomization and the first study medication. The eligible patients will be randomly assigned in a 5:1 ratio to receive 1 of 2 treatment groups in the treatment phase: Group 1: CNTO 136 10 mg/kg intravenous (IV), at Weeks 0, 4, 8, 12, 16, 20, 24; and Group 2: Placebo infusion, IV, at Weeks 0, 4, 8, 12, 16, 20, 24. Patients' medication regimen for LN may be adjusted from the Week 24 visit and afterwards. Safety evaluations for adverse events, infections, clinical laboratory tests, electrocardiogram, vital signs, physical examination and skin evaluations will be performed throughout the study. The follow up phase or the end of study will be the Week 40 visit for the last patient randomized, or, in the event that the last patient randomized withdraws from the study early, the end of study is defined as the date of the last visit of the last patient participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Systemic lupus erythematosus (SLE), and biopsy-proven International Society of Nephrology/Renal Pathology Society Class III or IV lupus glomerulonephritis within approximately 14 months prior to randomization
* Persistently active nephritis defined as, proteinuria greater than 0.5g/day as determined by measurement of total urine protein less than 0.5 g/24- hours or a urine Protein/Creatinine (P/C) ratio greater than 0.5 (mg/mg) in a timed collection of 12 or more hours, for 2 months or more prior to the first administration of study medication and observed during at least 2 visits conducted 1 week apart during the screening period
* Active Class III or Class IV lupus nephritis determined by recent biopsy within approximately 6 months prior to screening or at least 1 of the following 3 criteria: hematuria (blood in urine), anti-DNA positivity, or low C3 or C4 complement levels
* Stable immunosuppression for at least 9 weeks prior to the first administration of study medication consisting of MMF 1-3 g/day (or equivalent dose of MPA) with/without corticosteroids up to prednisone equivalent of 20 mg/day, or azathioprine 1-3 mg/kg/day with/without corticosteroids up to prednisone equivalent of 20 mg/day
* Stable dose of angiotensin-converting enzyme (ACE) inhibitor/angiotensin II receptor blocker (ARB) for at least 9 weeks prior to the first administration of study medication
* If using oral corticosteroids, must be on a stable dose equivalent to 20 mg/day or less of prednisone for at least 9 weeks prior to the first administration of study medication

Exclusion Criteria:

* Cyclophosphamide use within 3 months of randomization
* B-cell depletion therapy within 6 months of screening, or evidence of persistent B-cell depletion at the time of screening
* Greater than 50 percent glomerular sclerosis on renal biopsy
* Serum creatinine > 2.5 mg/dL (SI: > 177 µmol/L)
* White blood cell count < 3.5 x 10^3 cells/µL (SI: < 3.5 x 10^9 cells/L) or neutrophils < 1.96 x 10^3 cells/µL (SI: < 1.96 x 10^9 cells/L)
* Platelets < 140 x 103 cells/ µL (SI: < 140 x 10^9 cells/L)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with reduction in proteinuria (measurement of total urine protein greater than 0.5 g/24-hours, or a urine protein to creatinine ratio greater than 0.5 mg/mg) | Baseline to Week 24
  It is measured as the percentage in reduction of proteinuria from baseline to Week 24.

SECONDARY OUTCOMES:
Number of patients with a reduction from baseline in proteinuria by at least 50% | Up to Week 24
  It is measured as the proportion of patients with a reduction from baseline in proteinuria by at least 50% at any time through Week 24.
Number of patients with a meaningful reduction in proteinuria | Up to Week 24
  It is measured as the proportion of patients with meaningful reduction of proteinuria at any time through Week 24.
Number of patients with no worsening in Glomerular Filtration Rate (GFR) | Up to Week 24
  It is measured as the proportion of patients with no worsening in GFR at any time through Week 24.
Patient's Global Assessment of Disease Activity | Up to Week 24
  The Patient's Global Assessment of Disease Activity will be recorded on a visual analogue scale (VAS) (0 to 10 cm).
Physician's Global Assessment of Disease Activity | Up to Week 24
  The Physician's Global Assessment of Disease Activity will be recorded on a visual analogue scale (VAS) (0 to 10 cm).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (21):
- United States (8):
  - Birmingham, Alabama
  - Los Angeles, California
  - Chicago, Illinois
  - Lake Success, New York
  - Columbus, Ohio
  - Duncansville, Pennsylvania
  - Chattanooga, Tennessee
  - Carrollton, Texas
- Belgium (3):
  - Brussels
  - Leuven
  - Roeselare
- Mexico (4):
  - Guadalajara
  - Guadalajara, Jalisco
  - México
  - Querétaro
- Rotterdam, Netherlands
- Poland (3):
  - Gdansk
  - Warsaw
  - Wroclaw
- Thailand (2):
  - Bangkok
  - Chiang Mai

REFERENCES:
- [Derived] Rovin BH, van Vollenhoven RF, Aranow C, Wagner C, Gordon R, Zhuang Y, Belkowski S, Hsu B. A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Treatment With Sirukumab (CNTO 136) in Patients With Active Lupus Nephritis. Arthritis Rheumatol. 2016 Sep;68(9):2174-83. doi: 10.1002/art.39722. PMID 27110697